CLINICAL TRIAL: NCT04966897
Title: Randomized, Double-blind, Cross-over Trial Assessing a PERT-free Nutritional Therapeutic Delivery System for Cystic Fibrosis
Brief Title: Assessment of a PERT-free Nutritional Therapeutic Delivery System for Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlycosBio, Inc. (Industry)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GLYCOS-001-CF17
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: nutritional supplement; cystic fibrosis; PERT-free; pancreatic enzyme; enzyme modified oil; exocrine pancreatic insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, cross-over trial with a single blind stage evaluation assessing the GBNS for safety, tolerability and blood lipid levels compared to a standard nutritional supplement with PERT. Phase 1: After an overnight fast, subjects in Arm 1 administered PERT placebo with the GBNS and those in Arm 2 will be administered standard nutritional supplement with PERT. Blood samples collected at baseline and hourly over 6 hours for all subjects. Subjects will return for crossover treatment no fewer than 4 days and no more than 14 days after with the same steps as the above but with patients switching treatment arms. Phase 2: Starting the day following the 2nd treatment the 6 day, single-blind safety stage begins with subjects randomized to GBNS with PERT-placebo or the standard nutritional supplement with PERT. One week after the end of the Home Trial (+/- 3 days) patients will return for an end of study visit.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GBNS + PERT placebo (Experimental): GBNS + PERT placebo (drink volume sufficient to supply 0.5 g of MAG per kg of body weight plus PERT placebo capsules according to patient body weight.
  Interventions: Dietary Supplement: GlycosBio Nutritional Supplement + PERT placebo
- Standard Nutritional Supplement + PERT (Active Comparator): Standard nutritional supplement + PERT (drink volume sufficient to supply 0.5 g of TAG per kg of body weight plus PERT capsules according to body weight).
  Interventions: Dietary Supplement: Standard Nutritional Supplement + PERT

INTERVENTIONS:
Dietary Supplement: GlycosBio Nutritional Supplement + PERT placebo — The lipid (fat) in the GlycosBio Nutritional Supplement (GBNS) was provided in the form of a re-structured lipid monoacylglyceride (MAG) produced by the study sponsor. MAGs are readily absorbed by enterocytes without the need of digestion by pancreatic lipases. The "MAG oil" is produced enzymatically from almond oil. The product also contains essential amino acids, carbohydrates as simple sugars and fat-soluble vitamins and minerals. The GBNS to be administered in a volume sufficient to supply 0.5 g of MAG per kg of body weight
  Arms: GBNS + PERT placebo
Dietary Supplement: Standard Nutritional Supplement + PERT — A 5.9% fat triacylglycerol-based commercially available nutritional supplement (Boost Plus®, Nestlé Health Science, Bridgewater, NJ) in a volume sufficient to supply 0.5 g of TAG per kg of body weight over the same time period and PERT capsules (24,000 iu/capsule) at a dose of 2,500 iu of lipase activity per gram of fat ingested.
  Arms: Standard Nutritional Supplement + PERT

SUMMARY:
This is a single center, randomized, double-blind, cross-over trial (with a follow-on single-blind safety evaluation stage), assessing a ready-to-drink nutritional supplement used without PERT ("PERT-free"), nutritional supplement for blood lipid levels, safety and tolerability compared to a standard of care nutritional supplement used concomitantly with PERT.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, cross-over trial (with a follow-on single-blind safety evaluation stage), assessing a ready-to-drink nutritional supplement used without PERT ("PERT-free"), nutritional supplement for blood lipid levels, safety and tolerability compared to a standard of care nutritional supplement used concomitantly with PERT.

The study hypothesis is that the PERT-free nutritional supplement will be equivalent to, or superior to, a standardized nutritional shake with regard to fat absorption, as indicated by blood lipid (triglyceride) levels while maintaining tolerability and safety without the use of PERT. The objective is to evaluate efficacy, safety, and tolerability of a "PERT-free" nutritional shake compared to a standard nutritional shake used concomitantly with PERT. Measurements include components of a standard lipid blood panel (triglycerides, cholesterol, HDL cholesterol, LDL cholesterol, and VLDL cholesterol), absorption of fat-soluble vitamins (vitamin D) and symptoms associated with EPI. Other objectives include evaluating palatability and patients' impressions of the products.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 12 years or older.
* Diagnosis of cystic fibrosis
* Currently receiving treatment with a commercially available pancreatic enzyme product for more than 3 months.
* Clinically stable condition without evidence of acute respiratory disease within 1 month of enrollment.
* Stable body weight defined as no more than 5% decline within 3 months of enrollment.
* Females of child-bearing potential should agree to continue using a medically acceptable method of birth control throughout the study and for 30 days immediately after the last dose of study drug. Medically acceptable methods of birth control include bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection (Depo-Provera™), an intrauterine device, or an oral contraceptive taken within the past 3 months where the subject agrees to continue using during the study or to adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following: diaphragm, cervical cap, condom, or spermicide.
* Ability to take oral medication and oral liquid nutritional supplements and be willing to adhere to the study interventions.
* Agreement to adhere to Lifestyle Considerations as defined by the study protocol throughout the duration of the study.

Exclusion Criteria:

* Evidence of cardiovascular, respiratory (except underlying disease), urogenital, gastrointestinal/hepatic (except underlying disease), hematologic/immunologic, head, ears, eyes, nose, throat, dermatologic/connective tissue, musculoskeletal, metabolic/nutritional (except underlying disease), endocrine (except controlled diabetes mellitus), neurologic/psychiatric, milk, nut or soy allergies, recent major surgery, or other relevant diseases as revealed by history, physical examination and/or laboratory assessments, which could limit participation in or completion of the study.
* History of acute abdomen in the last year.
* History of fibrosing colonopathy.
* History of distal intestinal obstruction syndrome (DIOS) within 6 months prior to enrollment.
* Solid organ transplant or surgery affecting the large bowel other than appendectomy.
* Small bowel surgery that significantly affected absorptive capacity (e.g. gastrectomy or pancreatectomy).
* Intestinal inflammatory diseases including chronic diarrheal illness unrelated to pancreatic insufficiency.
* Celiac disease or Crohn's disease.
* Receiving enteral tube feeds for ≥50% of daily calorie intake.
* Pregnancy or lactation.
* Any type of malignancy involving the digestive tract in the last 5 years.
* Known allergy to pancreatin or inactive ingredients (excipients) of pancreatin capsules.
* Suspected non-compliance or non-cooperation.
* Intake of experimental drugs within 30 days prior to study start.
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subject's participation in or ability to complete the study.
* Diagnosis of human immunodeficiency virus in medical history.
* Listed for lung transplantation or other solid organ transplant or documented forced expiratory volume (FEV) ≤25%.
* Use of lipid lowering therapy including statins, fibrates, niacin, and proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitors that cannot be held at least 14 days prior to Day 1 and through Day 15 of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in serum triglyceride concentration | 6 hours
  Maximum change from baseline for serum triglyceride concentration based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
Maximum serum triglyceride concentration | 6 hours
  Maximum serum triglyceride concentration during the 6 hour period following administration of the oral nutritional supplement.
Area under the curve (AUC) for triglyceride serum levels | 6 hours
  Incremental area under the curve (AUC) for triglyceride serum levels during the 6 hour time period following following administration of the oral nutritional supplement.

SECONDARY OUTCOMES:
Serum glucose | 6 hours
  Maximum change from baseline for serum serum glucose based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
Total cholesterol | 6 hours
  Maximum change from baseline for serum total cholesterol based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
HDL cholesterol | 6 hours
  Maximum change from baseline for serum HDL cholesterol based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
LDL cholesterol | 6 hours
  Maximum change from baseline for serum LDL cholesterol based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
VLDL cholesterol | 6 hours
  Maximum change from baseline for serum VLDL cholesterol based on an hourly blood draw over a 6 hour period following administration of the oral nutritional supplement.
Incidence of gastrointestinal (GI) symptoms | 6 hours
  Incidence of gastrointestinal (GI) symptoms including nausea, heartburn, abdominal pain, steatorrhea, bloating and other reported symptoms over a 6 hour period following administration of the oral nutritional supplement.
Number of stools and other abdominal symptoms | 6 days
  Average daily number of stools and the percentage of days with 1) hard or formed/normal or soft stools, 2) no steatorrhea, 3) no abdominal pain, and 4) no bloating during the 6 days during Phase II (home phase) of trial.

OTHER OUTCOMES:
Palatability | 6 days
  Differences in the palatability of each oral nutritional supplement assessed via a participant survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center (CRC) at Texas Children's Hospital, Houston, Texas, United States